CLINICAL TRIAL: NCT07166029
Title: Effect of Russian Current on Hand Grip Strength and Functional Outcome After Carpal Tunnel Release
Acronym: CTS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Nawal Sayed Ahmed Ibrahim Ahmed, principle investigator : nawal sayed ahmed ibrahim ahmed, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P.T.REC/012/005964
Record Dates: First submitted 2025-09-03; First posted 2025-09-10 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Carpal Tunnel Syndrome
Keywords: carpal tunnel syndrome; russian current; hand grip strength
MeSH Terms: conditions — Carpal Tunnel Syndrome

STUDY DESIGN:
Intervention Model Description: russian current and tradional therapy
Who Masked: Outcomes Assessor
Masking Description: opaque sealed envelope
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- russian current (Experimental): 26 patients will receive Russian current plus a selected physical therapy program three times a week for four weeks.
  Interventions: Other: russian current; Other: selected physical therapy program
- selected physical therapy program (Active Comparator): 26 patients will receive a selected physical therapy program alone three times a week for four weeks.
  Interventions: Other: selected physical therapy program

INTERVENTIONS:
Other: russian current — russian current will be is applied in 50Hz sinusoidal bursts with a duty cycle of 50% (10ms on/10ms off). Russian Stimulation (at 2500Hz or 2.5kHz) has been shown to be effective in increasing muscle strength and torque generation through stimulation of type II muscle fiber. The stimulation will be given for duration of 10 minutes on followed by 50 sec off and again 10 sec on, three tims per week plus selsected physical therapy program.
  Arms: russian current
Other: selected physical therapy program — the patients will receive selected physical therapy program in the form of TENS for 15 min, US for 5 min and exercise for 20 min

SUMMARY:
this study will be conducted to investigate the effect of Russian current on hand grip strength and functional outcome after carpal tunnel release

DETAILED DESCRIPTION:
Carpal tunnel syndrome (CTS) is the most common entrapment neuropathy syndrome of the upper extremities , the estimated prevalence is 4-5% in the general population ,it occurs due to median nerve compression in carpal tunnel and it is ten times more common in women ,the most common symptoms are numbness and tingling in the radial 3-1/2 finger, night pain, and paresthesias. Although it is most commonly idiopathic, other causes include trauma, oral contraceptive use, pregnancy, arthritis, diabetes hypothyroidism, and repetitive wrist movements. It is well known that distal radius fractures and their sequelae can cause CTS, this suggests that anatomic changes in bony structures of wrist may also contribute to the development of CTS.Russian current (RC), a well-known neuromuscular electrical stimulation operating at 2500 Hz, has demonstrated significant strength improvement over traditional exercises due to its high tolerance and low pain provocation.There are studies about efficacy of Transcutaneous electrical nerve stimulation on wrist pain in patients with CTR but there is lack of literature about efficacy of RC on hand grip strength and function after CTR so this stidu will be conducted.

ELIGIBILITY:
Inclusion Criteria:

* Fifty-two patients with hand muscles weakness post operative carpal tunnel release ,due to severe carpal tunnel syndrome .
* Patient's age will range from 25 to 35 years.
* Patient's body mass index (BMI) will be less than 30kg/m2.
* Presence of wrist pain associated with hand grip weakness.

Exclusion Criteria:

* Patients with any other musculoskeletal or neurological disorders in the hand.
* Patients with a history of fractures and dislocations in the hand and wrist.
* Patients with hand deformities and edematous hands.
* Patients with cervical radiculopathy.
* Carpal tunnel syndrome due to conditions like hypothyroidism, rheumatoid arthritis, immunosuppression

Ages: 25 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 52 (Estimated)
Dates: Start 2025-09-15 (Estimated); Primary Completion 2025-11-30 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
hand grip strength | up to four weeks
  hand grip strength will be measured by hand held dynamometer.
fine and gross hand function | up to four weeks
  jebsen taylor hand test will be used to assess fine and gross hand function.this test includes series of seven subtests representing fine motor, nonweighted and weighted hand function in ADL, which includes printing a 24-letter, third-grade reading difficulty sentence, Turning over 7.6×12.7 cm (3×5-inch) cards (simulated page turning), Picking up small, common objects (e.g. pennies, paper clips, bottle caps) and placing them in a container,Stacking checkers (test of eye-hand co-ordination),Simulated feeding, Moving large empty cans, Moving large weighted [0.45 kg (l lb)] cans.The subtests are scored by recording the number of seconds required to complete each test
hand function | up to four weeks
  hand function will be measured by boston carpal tunnel questionnaire.The Boston Carpal Tunnel Questionnaire (BCTQ) is a patient-reported questionnaire used to assess symptoms and functional limitations in people with carpal tunnel syndrome (CTS). It consists of two modules: an 11-item Symptom Severity Scale (SSS) and an 8-item Functional Status Scale (FSS), which are scored independently on a 1-to-5 Likert scale.A mean score between 1 and 5 is generated for both the SSS and FSS, with higher scores indicating more severe symptoms or greater functional limitation.

SECONDARY OUTCOMES:
wrist range of motion | up to four weeks
  goniometer device will be used to assess wrist range of motion
pain intensity | up to four weeks
  pain will be measured by visual analogue scale. Scores are based on self-reported measures of symptoms that are recorded with a single handwritten mark placed at one point along the length of a 10-cm line that represents a continuum between the two ends of the scale-"no pain" on the left end (0 cm) of the scale and the "worst pain" on the right end of the scale (10 cm).